CLINICAL TRIAL: NCT05516186
Title: Effects of a Scapular-focused Exercise Protocol for Patients With Rotator Cuff Related Pain Syndrome - a Randomized Clinical Trial
Brief Title: Effects of a Scapular-focused Exercise Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NOVA School of Science and Technology ı FCT NOVA (Other)
Responsible Party: Principal Investigator, Ricardo Matias, PhD, NOVA School of Science and Technology ı FCT NOVA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/2022 ESSAlcoitão
Record Dates: First submitted 2022-08-11; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Rotator Cuff Syndrome of Shoulder and Allied Disorders
Keywords: scapula neuromuscular activity and control; rotator cuff related pain syndrome; scapular dyskinesis; electromyographic biofeedback; control therapy; pain and function
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scapular-focused exercise protocol supported by real-time EMGBF (Experimental): The scapular-focused exercise protocol followed the protocol described by dos Santos et al. (2021). The protocol uses sequential stages of motor relearning (cognitive, associative, and autonomous) as a framework, while promoting the integration of local and global muscle function in weekly sessions divided into three phases. The main purpose of the protocol is to increase scapular neuromuscular activity and control.
  Interventions: Other: Control Therapy; Other: Scapular-focused exercise protocol without EMGBF
- Scapular-focused exercise protocol without EMGBF (Experimental): The same protocol described above was applied without EMGBF
  Interventions: Other: Scapular-focused exercise protocol with EMGBF; Other: Control Therapy
- Control therapy group (Other): The control therapy group underwent conservative physical therapy, which included both manual and exercise therapy
  Interventions: Other: Scapular-focused exercise protocol with EMGBF; Other: Scapular-focused exercise protocol without EMGBF

INTERVENTIONS:
Other: Scapular-focused exercise protocol with EMGBF — Scapular-focused exercises, based on the dos Santos et al (2021) protocol with the aid of the electromyographic biofeedback
  Arms: Control therapy group; Scapular-focused exercise protocol without EMGBF
Other: Control Therapy — manual and exercise therapy
  Arms: Scapular-focused exercise protocol supported by real-time EMGBF; Scapular-focused exercise protocol without EMGBF
Other: Scapular-focused exercise protocol without EMGBF — Scapular-focused exercises, based on the dos Santos et al (2021) protocol
  Arms: Control therapy group; Scapular-focused exercise protocol supported by real-time EMGBF

SUMMARY:
Background: Current clinical practice still lacks consistent evidence in the physiotherapy management of Rotator cuff related pain syndrome (RCS). The purpose of this trial was to compare the effectiveness of a scapular-focused treatment with and without real-time electromyographic biofeedback (EMGBF) to a control therapy in patients with RCS.

Methods: 60 patients with RCS were divided into three groups: scapular-focused exercise protocol group (P_G n=20), scapular-focused exercise protocol with EMGBF group (P+EMGBF_G n=20) and control therapy group (CT_G n=20). Values of pain and function [Shoulder Pain and Disability Index (SPADI) questionnaire, complemented by the Numeric Pain Rating Scale (NPRS) and Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire], scapular stabilizer neuromuscular control (SSNC), scapular stabilizer activation onset (SSAO), dynamic scapular alignment, range of motion (ROM) and glenohumeral flexor and abductor muscle strength (GMS) were assessed at baseline and after 6-weeks and compared within and between groups.

DETAILED DESCRIPTION:
In order to advance the understanding of the value of scapular-focused exercise for rotator cuff related syndrome, a new trial was designed with the main objective of comparing pain and function outcomes between three different treatment protocols for patients with RCS:

P_G - Scapular-focused exercise protocol without electromyographic biofeedback (EMGBF) P+EMGBF_G - Scapular-focused exercise protocol supported by real-time EMGBF CT_G - Control therapy group with manual therapy (glenohumeral joint physiologic and accessory mobilization) , massage to reduce upper trapezius (UT) stiffness, and shoulder rotation strengthening into external rotation Every outcomes was assessed at the beginning of treatment, and then, weekly until completed 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1- age between 18 and 60 years; 2 - primary complaint of shoulder pain 3 - RCS clinical diagnosis

Exclusion Criteria:

1. - neurological symptoms;
2. - positive thoracic outlet syndrome (screened with Allen's and Adson's tests);
3. - history of shoulder surgery or fracture;
4. - structural injuries confirmed by imaging (e.g. ligaments and labrum);
5. - symptoms reproduced by cervical examination;
6. - unable to commit to scheduled treatments;
7. - Anti-inflammatory drug use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
NPRS numeric pain rating scale | At the initial assessment
  From zero (better score) to 10 (worst score)
NPRS numeric pain rating scale | At 6 weeks after the treatment protocol (final assessment)
  From zero (better score) to 10 (worst score)
SPADI shoulder pain and disability index | At the initial assessment
  From zero (better score) to 100 (worst score)
SPADI shoulder pain and disability index | At 6 weeks after the treatment protocol (final assessment)
  From zero (better score) to 100 (worst score)
DASH disabilities of the arm, shoulder and hand | At the initial assessment
  From zero (better score) to 100 (worst score)
DASH disabilities of the arm, shoulder and hand | At 6 weeks after the treatment protocol (final assessment)
  From zero (better score) to 100 (worst score)

SECONDARY OUTCOMES:
scapular stabilizer neuromuscular control | At the initial assessment
  Electromyographic Biofeedback (EMGBF) PhysiopluxTM system version 1.06
scapular stabilizer neuromuscular control | At 6 weeks after the treatment protocol (final assessment)
  Electromyographic Biofeedback (EMGBF) PhysiopluxTM system version 1.06
scapular stabilizer activation onset | At the initial assessment
  Electromyographic Biofeedback (EMGBF) PhysiopluxTM system version 1.06
scapular stabilizer activation onset | At 6 weeks after the treatment protocol (final assessment)
  Electromyographic Biofeedback (EMGBF) PhysiopluxTM system version 1.06
dynamic scapular alignment | At the initial assessment
  Observation of the medial and the inferior prominences of the scapula
dynamic scapular alignment | At 6 weeks after the treatment protocol (final assessment)
  Observation of the medial and the inferior prominences of the scapula
range of motion | At the initial assessment
  Goniometry
range of motion | At 6 weeks after the treatment protocol (final assessment)
  Goniometry
glenohumeral flexor and abductor muscle strength | At the initial assessment
  Manual Testing From 0 (worst) to 5 (normal)
glenohumeral flexor and abductor muscle strength | At 6 weeks after the treatment protocol (final assessment)
  Manual Testing From 0 (worst) to 5 (normal)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Almeida, MsC, Study Chair — Superior School of Health os Setúbal
Locations (1):
- Policlínica de Sátão, Viseu, Portugal

IPD SHARING:
Plan to Share IPD: No